CLINICAL TRIAL: NCT02757599
Title: Impact of Image Orientation During Transvaginal Ultrasound on Learning: A Randomized Trial
Brief Title: Top-down Versus Bottom-up Transvaginal Ultrasound Scan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Caroline Amalie Taksoe-Vester, Stud.med, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12345
Record Dates: First submitted 2016-04-18; First posted 2016-05-02 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Transvaginal Ultrasound Scan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Top-down (TD) (Other): The group having the transvaginal ultrasound image top-down. During training and transfer test.
  Interventions: Other: Ultrasound training
- Bottom-up (BU) (Other): The group having the transvaginal ultrasound image bottom-up. During training and transfer test.
  Interventions: Other: Ultrasound training

INTERVENTIONS:
Other: Ultrasound training — Training on the transvaginal ultrasound simulator.

SUMMARY:
Background: Transvaginal ultrasound training of novices is performed differently with respect to the orientation of the ultrasound image. There is no international consensus on the orientation of the transvaginal ultrasound image and no evidence to support whether one orientation is superior to the other in terms of educational outcome and learning curves.

The aim of this study is to assess the effects of transvaginal ultrasound training when orienting the image top-down versus bottom-up, which can open for the discussion concerning a uniform transvaginal ultrasound education. This study may improve ultrasound novices' learning and potentially ensure that future clinicians perform transvaginal ultrasound examinations in the same manner.

Hypotheses: The investigators hypothesize that the orientation perceived by ultrasound novices, as the most intuitive will result in lower cognitive load during training and result in shorter learning curves and improved transfer of skills to various settings and cases.

DETAILED DESCRIPTION:
Background

Ultrasonography is considered safe but highly operator dependent. Ultrasonography is being used increasingly in gynecology and obstetrics; however the training of novices in transvaginal ultrasound is performed differently with respect to the orientation of the ultrasound image, which often differs between operators and institutions. The image may be oriented top- down (transducer at the top) or bottom-up (transducer at the bottom). The different orientations of the image are a challenge for novices when being supervised by senior clinicians with different preferences for image orientation. As for now, there is no international consensus on image orientation and there is no evidence to support the superiority of one over the other in terms of learning curves and educational outcomes such as skills transfer. Transvaginal ultrasound is, like all other kinds of ultrasound, associated with long learning curves and is therefore time-consuming and requires extensive training. Transvaginal ultrasound is often associated with some discomfort to the patient, which can be reduced with adequate initial training. It therefore seems reasonable to determine how to provide the most effective initial transvaginal ultrasound training to reduce unnecessary patient discomfort and improve diagnostic accuracy through accelerated learning curves.

A recent study involving laparoscopic training, suggests that novices learn best from simplified practice during initial skills acquisition because it allows them to deal with future task complexity better than when being faced with complex image orientation. These findings are consistent with cognitive load theory, which emphasizes the limitations of the working memory when learning new tasks. Optimal learning occurs when the cognitive load of a new task is within the limits of the learner's working memory and when instructional features that do not contribute to learning are eliminated. Basic knobology (operating the ultrasound machine controls) and image interpretation represent significant sources of cognitive load for ultrasound novices and the acquisition of images should therefore be as simple as possible to avoid exceeding the working memory of the learner.

When looking at an ultrasound image, the operator transforms the two-dimensional ultrasound image into a three-dimensional internal representation of the structure being examined. Alignment of the image according to the physical angle of the transvaginal ultrasound probe by having the image facing bottom-up is by some clinicians perceived as the most intuitive anatomical orientation. Other clinicians prefer having the ultrasound image oriented the same way (top-down) regardless of the type of examination being performed (transabdominal or transvaginal).

The research question in this study is:

In a group of ultrasound novices, what is the effect of the transvaginal ultrasound training when orienting the image top-down versus bottom-up on learning curves and transfer of skills to different settings and cases?

Hypotheses:

The investigators hypothesize that the orientation perceived by ultrasound novices as the most intuitive will also result in shorter learning curves and improved transfer of skills. This study may improve ultrasound novices' learning and ensure that future clinicians perform transvaginal ultrasound examinations in the same manner. If the orientation of the image does not result in any changes to educational outcomes, there is no argument for adopting one approach over the other from an educational point-of-view.

Participants

Participants in this study are medical students from the University of Copenhagen, Denmark. Inclusion criteria require that participants 1) are medical students from year 3 to year 6; 2) have no previous ultrasound experience besides a mandatory ultrasound course of four hours provided at the 6th semester for medical students at the University of Copenhagen; and 3) provide written informed consent. Participants are after inclusion randomly divided into two study groups:

1. Group one (TD): Orienting the transvaginal ultrasound image top-down
2. Group two (BU): Orienting the transvaginal ultrasound image bottom-up

Randomization An independent research fellow at the Copenhagen Academy for Medical Education and Simulation, Rigshospitalet, randomizes participants by computer to either of the two groups.

Intervention Before any training is commenced, all participants are surveyed on their intuitive preferences for image orientation. Participants in both groups then receive a short theoretical introduction to pelvic ultrasound. Afterwards the participants are introduced to the simulated environment and the Virtual Reality (VR) simulator (Scantrainer) used for training. The VR simulator provides images obtained from real patients and haptic feedback from the ultrasound probe.

The study is based on the principle of mastery learning, thus participants are instructed to complete a simulator test that includes a number of practice modules until they have reached expert levels of performance. The expert performance level has been established in a previous validation study. Participants in the TD and BU groups are instructed with the ultrasound image top-down and bottom-up, respectively, throughout all training and assessment.

When the expert level is reached the participants perform a transfer test on the low-fidelity simulator (BluePhantom) within 7 days of completed simulator training. During the transfer test participants will be asked to complete a systematic ultrasound examination and to optimize the images during the scan. The performances will be videotaped and afterwards rated by two clinicians used to perform transvaginal ultrasound - one clinician used to seeing the ultrasound image top-down and the other clinician used to seeing the image bottom-up. The participants will be rated using the Objective Structured Assessment of Ultrasound Skills.

After completed training, participants are assessed on their cognitive load using a cognitive load questionnaire.

All training and assessments take place in the simulated setting in the skills lab at Copenhagen Academy for Medical Education and Simulation, Rigshospitalet.

Outcomes

Primary outcome:

• The primary outcome measures include learning curve for the two groups and performances during the transfer test. Learning curves are assessed through simulator scores obtained on the practice modules. A previous study has demonstrated that mastery learning levels are attained after four to five rounds of training on the practice modules included in the simulator test

Secondary outcomes:

* Participants' perception of the most intuitive approach before training.
* Time used within the two groups to reach expert level
* Cognitive load measurements using the instrument described by Leppink et al. after training

ELIGIBILITY:
Inclusion Criteria:

1. are medical students from year 3 to year 6
2. provide written informed consent.

Exclusion Criteria:

1) Have previous ultrasound experience besides a mandatory ultrasound course of four hours provided at the 6th semester for medical students at the University of Copenhagen

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Learning curve measured by time used for training | 6 months

SECONDARY OUTCOMES:
Cognitive load, measured by a questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline A Taksoe-Vester, Bach.med, Principal Investigator — Student teacher

IPD SHARING:
Plan to Share IPD: Yes